CLINICAL TRIAL: NCT02438137
Title: A Randomized Clinical Trial of Dimethyl Fumarate as a Novel Therapeutic Agent for Obstructive Sleep Apnea
Brief Title: Dimethyl Fumarate for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tiffany J. Braley, MD, MS, Assistant Professor, Department of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00080121
Record Dates: First submitted 2015-04-18; First posted 2015-05-08 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea; OSA; Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; sleep apnea; snoring; dimethyl fumarate; CPAP; continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dimethyl Fumarate (Tecfidera®) capsules (Active Comparator): The starting dose for dimethyl fumarate (Tecfidera®, http://www.tecfidera.com/pdfs/full-prescribing-information.pdf) is 120 mg twice a day orally. After 7 days, the dose should be increased to the maintenance dose of 240 mg twice a day, though slower dose escalations are possible to increase tolerability, if necessary. Participants randomized to dimethyl fumarate will be instructed to take this medication twice a day with breakfast and dinner for a period of 4 months.
  Interventions: Drug: Dimethyl fumarate
- Placebo (Placebo Comparator): The placebo is an inert product that looks like a pill and is identical to dimethyl fumarate capsules, but it contains no medicine. Participants randomized to placebo will be instructed to take placebo twice a day with breakfast and dinner for a period of 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl fumarate — Dimethyl fumarate capsules will be dispensed during routine study appointments. 120 mg tablets will be dispensed to facilitate dose titrations. Drug will be dispensed in 1 month supply, so that compliance can be reconciled at monthly follow-up visits, and recorded in accountability logs. Participants will be instructed to take the medication with food, in the morning and at dinnertime. If participants miss a dose, they will be instructed to resume their normal dose at the next scheduled time, and be instructed not to take an extra dose at their next dosing interval if they previously miss a dose.
  Other Names: Tecfidera
  Arms: Dimethyl Fumarate (Tecfidera®) capsules
Drug: Placebo — Placebo capsules will be dispensed during routine study appointments. Placebo will be dispensed in 1 month supply, so that compliance can be reconciled at monthly follow-up visits, and recorded in accountability logs. Participants will be instructed to take the placebo with food, in the morning and at dinnertime. If participants miss a dose, they will be instructed to resume their normal dose at the next scheduled time, and be instructed not to take an extra dose at their next dosing interval if they previously miss a dose.
  Arms: Placebo

SUMMARY:
The overall purpose of this study is to determine whether the oral medication dimethyl fumarate is an effective treatment for obstructive sleep apnea in patients who are unable, unwilling, or uneager to use positive airway pressure therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder that involves collapse of the upper airway during sleep, leading to low blood oxygen levels and sleep disruption. Untreated OSA increases the risk of many health consequences, including high blood pressure, heart disease, stroke, diabetes, memory problems, fatigue, sleepiness, and impaired memory. Despite its profound public health and societal impact, there are no known medications that can effectively treat OSA, and up to 50% of patients cannot tolerate current treatments. The primary treatment for OSA, known as Continuous Positive Airway Pressure (CPAP), is delivered by a mechanical device and mask that blows air into the airway to keep it open during sleep. Although CPAP controls OSA, many patients can't tolerate the discomfort of the mask, and up to 50% of patients cannot use CPAP appropriately.

Several recent studies of OSA patients suggest that inflammation in the airway and the bloodstream may worsen OSA, and that medications that control inflammation may improve OSA. In particular, a previous study from the researchers suggests that multiple sclerosis (MS) patients who are on MS therapies that control inflammation may have less severe OSA than those who are not. MS is an autoimmune disease that is associated with inflammation of the nervous system. As OSA may also be caused or worsened by inflammation, this clinical trial aims to study the effects of a specific MS medication known as dimethyl fumarate (brand name - Tecfidera®) to see if it may also be useful to treat OSA. Tecfidera® is already approved by the Food and Drug Administration (FDA) to treat patients with MS. However, it is not approved by the FDA for the treatment of OSA and is thus considered an investigational drug in this study.

Study-related activities will last for 5 months. Consenting participants will receive a baseline overnight sleep study to assess their current sleep apnea severity. Participants will then be given either oral dimethyl fumarate or placebo for a period of 4 months, and will be followed on a monthly basis during the course of the study. At the end of the study, participants will undergo a repeat overnight sleep study to monitor for changes in their sleep apnea severity. Treatments will be assigned at random (like flipping a coin), and participants will not be aware of which treatment they receive. There is a 2/3 chance that participants will receive dimethyl fumarate. Participants will also undergo blood draws and complete several surveys during their monthly study visits. Participants will be compensated for their travel and time throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years at screening;
2. Diagnosis of OSA as confirmed by previous clinical sleep study (polysomnography, PSG);
3. Refusal, inability, or high reluctance to use CPAP regularly for treatment of OSA, despite medical advice;
4. Willingness to undergo repeat sleep study (PSG) and blood studies;
5. Normal immune cell counts, as evidenced by complete blood count (CBC) done at screening

Exclusion Criteria:

1. Regular use of CPAP within the last 2 months
2. Physical, psychiatric or cognitive impairment that prevents informed consent, PSG, or reliable follow-up;
3. Cardiac conditions that may increase sleep apnea severity (e.g., congestive heart failure or recent heart attack);
4. Current successful treatment for obstructive or central sleep apnea, for example by CPAP, and patient agreement to continue with that treatment;
5. History of surgical treatment for OSA within past 6 months, or subsequent to last PSG confirmation that OSA is present;
6. Active nervous system diseases that may predispose subjects to OSA;
7. Systemic autoimmune disease that could increase inflammation and influence apnea severity (such as rheumatoid arthritis or lupus);
8. Pregnancy or breastfeeding;
9. Use of immunotherapies or immunosuppressants, currently or within past 6 months;
10. Anticipated initiation or dose change in tricyclic antidepressants, selective serotonin uptake inhibitors, or related compounds;
11. Participants with a history of active, serious or persistent infections.
12. Participants with recent surgery (within 3 months prior to screening), or anticipated surgery during the length of the study.
13. Systemic steroid use within the last 2 months (does not include local steroid injections or intranasal steroid spray);
14. Current diagnosis of cancer that is not considered to be cured or in remission by the treating physician, cancer treatment of any kind within the last 6 months prior to screening (chemo, radiation, surgery), or anticipated cancer treatment during the length of the study;
15. History of a lymphoproliferative disorder (such as leukemia);
16. History of Multiple Myeloma
17. History of decreased immune cell counts per a blood test known as a CBC, specifically lymphocyte counts less than 1.2 K/μL at screening.
18. Refusal to use at least one reliable method of birth control (for women of childbearing age)
19. Newly diagnosed (within 2 months) OSA subjects who have an AHI > 30 and history of serious, recent, or unstable cardiovascular disease (including but not limited to recent MI, recent stroke/TIA, or unstable angina)
20. Participants who report previous motor vehicle accidents or near-misses presumed to be due to excessive sleepiness while driving.
21. Any other condition or treatment that in the opinion of the investigator could affect subject safety or study eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany J. Braley, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aloia MS, Stanchina M, Arnedt JT, Malhotra A, Millman RP. Treatment adherence and outcomes in flexible vs standard continuous positive airway pressure therapy. Chest. 2005 Jun;127(6):2085-93. doi: 10.1378/chest.127.6.2085. PMID 15947324
- [Background] Vgontzas AN, Bixler EO, Tan TL, Kantner D, Martin LF, Kales A. Obesity without sleep apnea is associated with daytime sleepiness. Arch Intern Med. 1998 Jun 22;158(12):1333-7. doi: 10.1001/archinte.158.12.1333. PMID 9645828
- [Background] Vgontzas AN, Zoumakis E, Lin HM, Bixler EO, Trakada G, Chrousos GP. Marked decrease in sleepiness in patients with sleep apnea by etanercept, a tumor necrosis factor-alpha antagonist. J Clin Endocrinol Metab. 2004 Sep;89(9):4409-13. doi: 10.1210/jc.2003-031929. PMID 15356039
- [Background] Thomas KS, Motivala S, Olmstead R, Irwin MR. Sleep depth and fatigue: role of cellular inflammatory activation. Brain Behav Immun. 2011 Jan;25(1):53-8. doi: 10.1016/j.bbi.2010.07.245. Epub 2010 Jul 23. PMID 20656013
- [Background] Aihara K, Oga T, Chihara Y, Harada Y, Tanizawa K, Handa T, Hitomi T, Uno K, Mishima M, Chin K. Analysis of systemic and airway inflammation in obstructive sleep apnea. Sleep Breath. 2013 May;17(2):597-604. doi: 10.1007/s11325-012-0726-y. Epub 2012 Jun 7. PMID 22674397
- [Background] Tam CS, Wong M, McBain R, Bailey S, Waters KA. Inflammatory measures in children with obstructive sleep apnoea. J Paediatr Child Health. 2006 May;42(5):277-82. doi: 10.1111/j.1440-1754.2006.00854.x. PMID 16712558
- [Background] Ursavas A, Karadag M, Rodoplu E, Yilmaztepe A, Oral HB, Gozu RO. Circulating ICAM-1 and VCAM-1 levels in patients with obstructive sleep apnea syndrome. Respiration. 2007;74(5):525-32. doi: 10.1159/000097770. Epub 2006 Dec 4. PMID 17148932
- [Background] Cofta S, Wysocka E, Dziegielewska-Gesiak S, Michalak S, Piorunek T, Batura-Gabryel H, Torlinski L. Plasma selectins in patients with obstructive sleep apnea. Adv Exp Med Biol. 2013;756:113-9. doi: 10.1007/978-94-007-4549-0_15. PMID 22836626
- [Background] Htoo AK, Greenberg H, Tongia S, Chen G, Henderson T, Wilson D, Liu SF. Activation of nuclear factor kappaB in obstructive sleep apnea: a pathway leading to systemic inflammation. Sleep Breath. 2006 Mar;10(1):43-50. doi: 10.1007/s11325-005-0046-6. PMID 16491391
- [Background] Walsh JA, Duffin KC, Crim J, Clegg DO. Lower frequency of obstructive sleep apnea in spondyloarthritis patients taking TNF-inhibitors. J Clin Sleep Med. 2012 Dec 15;8(6):643-8. doi: 10.5664/jcsm.2254. PMID 23243397
- [Background] Braley TJ, Segal BM, Chervin RD. Sleep-disordered breathing in multiple sclerosis. Neurology. 2012 Aug 28;79(9):929-36. doi: 10.1212/WNL.0b013e318266fa9d. Epub 2012 Aug 15. PMID 22895593
- [Background] Gerdes S, Shakery K, Mrowietz U. Dimethylfumarate inhibits nuclear binding of nuclear factor kappaB but not of nuclear factor of activated T cells and CCAAT/enhancer binding protein beta in activated human T cells. Br J Dermatol. 2007 May;156(5):838-42. doi: 10.1111/j.1365-2133.2007.07779.x. Epub 2007 Mar 23. PMID 17381463
- [Background] Stoof TJ, Flier J, Sampat S, Nieboer C, Tensen CP, Boorsma DM. The antipsoriatic drug dimethylfumarate strongly suppresses chemokine production in human keratinocytes and peripheral blood mononuclear cells. Br J Dermatol. 2001 Jun;144(6):1114-20. doi: 10.1046/j.1365-2133.2001.04220.x. PMID 11422029
- [Background] Wierinckx A, Breve J, Mercier D, Schultzberg M, Drukarch B, Van Dam AM. Detoxication enzyme inducers modify cytokine production in rat mixed glial cells. J Neuroimmunol. 2005 Sep;166(1-2):132-43. doi: 10.1016/j.jneuroim.2005.05.013. PMID 15993952
- [Background] Vandermeeren M, Janssens S, Borgers M, Geysen J. Dimethylfumarate is an inhibitor of cytokine-induced E-selectin, VCAM-1, and ICAM-1 expression in human endothelial cells. Biochem Biophys Res Commun. 1997 May 8;234(1):19-23. doi: 10.1006/bbrc.1997.6570. PMID 9168952
- [Background] Wallbrecht K, Drick N, Hund AC, Schon MP. Downregulation of endothelial adhesion molecules by dimethylfumarate, but not monomethylfumarate, and impairment of dynamic lymphocyte-endothelial cell interactions. Exp Dermatol. 2011 Dec;20(12):980-5. doi: 10.1111/j.1600-0625.2011.01376.x. Epub 2011 Oct 13. PMID 21995308
- [Background] Meissner M, Valesky EM, Kippenberger S, Kaufmann R. Dimethyl fumarate - only an anti-psoriatic medication? J Dtsch Dermatol Ges. 2012 Nov;10(11):793-801. doi: 10.1111/j.1610-0387.2012.07996.x. Epub 2012 Aug 17. English, German. PMID 22897153
- [Background] Scannevin RH, Chollate S, Jung MY, Shackett M, Patel H, Bista P, Zeng W, Ryan S, Yamamoto M, Lukashev M, Rhodes KJ. Fumarates promote cytoprotection of central nervous system cells against oxidative stress via the nuclear factor (erythroid-derived 2)-like 2 pathway. J Pharmacol Exp Ther. 2012 Apr;341(1):274-84. doi: 10.1124/jpet.111.190132. Epub 2012 Jan 20. PMID 22267202
- [Derived] Braley TJ, Huber AK, Segal BM, Kaplish N, Saban R, Washnock-Schmid JM, Chervin RD. A randomized, subject and rater-blinded, placebo-controlled trial of dimethyl fumarate for obstructive sleep apnea. Sleep. 2018 Aug 1;41(8). doi: 10.1093/sleep/zsy109. PMID 29800466

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimethyl Fumarate (Tecfidera®) Capsules: The starting dose for dimethyl fumarate was 120 mg twice a day orally. After 7 days, the dose was increased to the maintenance dose of 240 mg twice a day. Slower dose escalations were allowed to increase tolerability, if necessary. Participants randomized to dimethyl fumarate were instructed to take this medication twice a day with breakfast and dinner for a period of 4 months.
  Dimethyl fumarate: Dimethyl fumarate capsules were dispensed at routine study appointments. 120 mg tablets were dispensed to facilitate dose titrations. Drug was dispensed in 1 month supply, so that compliance could be reconciled at follow-up visits, and recorded in accountability logs. Participants were instructed to take medication with food, (morning and at dinnertime). If participants missed a dose, they were instructed to resume their normal dose at the next scheduled time, and not to take an extra dose at their next dosing interval if they previously miss a dose.
- Placebo: The placebo is an inert product that looks like a pill and is identical to dimethyl fumarate capsules, but it contains no medicine. Participants randomized to placebo were instructed to take placebo twice a day with breakfast and dinner for a period of 4 months.
  Placebo: Placebo capsules were dispensed during routine study appointments. Placebo were dispensed in 1 month supply, so that compliance could be reconciled at monthly follow-up visits, and recorded in accountability logs. Participants were instructed to take the placebo with food, in the morning and at dinnertime. If participants missed a dose, they were instructed to resume their normal dose at the next scheduled time, and not to take an extra dose at their next dosing interval if they previously missed a dose.
Period: Overall Study
Arm/Group | Dimethyl Fumarate (Tecfidera®) Capsules | Placebo
Started | 44 | 21
Completed | 36 | 15
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 65 participants were randomized and included in baseline analyses. 14 participants withdrew from the study or were lost to followup. 51 participants completed study activities. 50 participants (35 DMF and 15 placebo) who both completed the study and had an interpretable Month 4 PSG were included in the final analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dimethyl Fumarate (Tecfidera®) Capsules | Placebo | Total
Number analyzed (Participants) | 44 | 21 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.7) | 52.5 (12.4) | 50.2 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 20 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 44 | 21 | 65
Respiratory Disturbance Index (RDI) [Mean (Standard Deviation); unit: respiratory events/hour] — The RDI represents the total number of apneas, hypopneas and respiratory-related arousals per hour of sleep.
  respiratory events/hour | 36.4 (28) | 29.0 (16.9) | 34 (25.1)
Baseline cytokine levels (log-transformed values) [Mean (Standard Deviation); unit: pg/ml]
  Interleukin-6 | 0.406 (0.354) | 0.300 (0.249) | 0.372 (0.325)
  Tissue Necrosis Factor-alpha | 0.933 (0.195) | 1.009 (0.354) | 0.957 (0.257)
  Interleukin-10 | 0.596 (0.558) | 0.392 (0.294) | 0.530 (0.496)
  Monocyte Chemoattractant Protein-1 | 2.632 (0.118) | 2.593 (0.210) | 2.619 (0.153)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Apnea Severity as Measured by the Respiratory Disturbance Index (RDI)
Description: For the 50 participants who had interpretable month 4 polysomnography (PSG) data available, mean change in sleep apnea severity, as measured by the mean change in respiratory disturbance index (RDI) between baseline (Month 0) PSG and Month 4 PSG, was calculated. The RDI represents the total number of apneas, hypopneas and respiratory-related arousals per hour of sleep.
Time Frame: Month 0 to Month 4
Population: 65 participants were randomized. 14 participants withdrew from the study or were lost to followup. 51 completed study activities. 50 (35 DMF and 15 placebo) both completed the study and had an interpretable Month 4 PSG. One participant's Month 4 PSG was uninterpretable, thus the RDI from this participant could not be included in the final analysis.
Measure: Mean (Standard Deviation); unit: respiratory events/hour
Groups:
- Placebo: The placebo is an inert product that looks like a pill and is identical to dimethyl fumarate capsules, but it contains no medicine. Participants randomized to placebo will be instructed to take placebo twice a day with breakfast and dinner for a period of 4 months.
  Placebo: Placebo capsules were dispensed during routine study appointments. Placebo were dispensed in 1 month supply, so that compliance can be reconciled at monthly follow-up visits, and recorded in accountability logs. Participants were instructed to take the placebo with food, in the morning and at dinnertime. If participants missed a dose, they were instructed to resume their normal dose at the next scheduled time, and not to take an extra dose at their next dosing interval if they previously missed a dose.
Arm/Group | Dimethyl Fumarate (Tecfidera®) Capsules | Placebo
Number analyzed (Participants) | 35 | 15
respiratory events/hour | -3.11 (12.9) | 10.2 (13.1)
Statistical Analysis 1: Comparison: Dimethyl Fumarate (Tecfidera®) Capsules vs Placebo; Multiple linear regression models were used to calculate treatment effect (DMF or placebo) on mean RDI change, controlling for change in age, gender, BMI, time spent in supine sleep, and time spent in REM sleep; Test type: Superiority — In multiple linear regression models, the effect of DMF treatment on mean RDI change (beta-coefficient) was -11.3 respiratory events per hour (p=0.0124); p = 0.0124, Regression, Linear; beta-coefficient for treatment effect = -11.3, Standard Error of Mean 4.3; A mixed effects model, which treated RDI as a repeated measure and used individual ID as random effect, adjusted for age, gender, BMI, time spent in supine sleep, was also conducted. In this model, the effect of DMF compared to placebo, controlling for all other covariates, is a 28% decrease in Month 4 RDI (p=0.033)

2. Secondary Outcome: Mean Change in Serum Cytokine Levels (Mean Difference of Log-transformed Values)
Description: Levels of markers in the blood known as cytokines (measured in picograms per milliliter) were measured on a monthly basis from Month 0 (baseline) to Month 4. The outcome is the mean difference in cytokine level from baseline to month 4 (mean level at Month 4 - mean level at Baseline). Values were log-transformed for normality, prior to analysis.
Time Frame: Month 0 to Month 4
Population: Cytokine analyses were conducted for those participants who completed the study and had interpretable Month 4 PSG results. Among this group, 3 participants did not have usable Month 4 blood specimens for this analysis. Thus, the mean difference in cytokine levels was calculated for 47 participants.
Measure: Mean (Standard Deviation); unit: picograms/milliliter (log-transformed)
Groups:
- Dimethyl Fumarate (Tecfidera®) Capsules: The starting dose for dimethyl fumarate was 120 mg twice a day orally. After 7 days, the dose was increased to the maintenance dose of 240 mg twice a day, though slower dose escalations were possible to increase tolerability, if necessary. Subjects randomized to dimethyl fumarate were instructed to take this medication twice a day with breakfast and dinner for a period of 4 months.
  Dimethyl fumarate: Dimethyl fumarate capsules were dispensed at routine study appointments. 120 mg tablets were dispensed to facilitate dose titrations. Drug was dispensed in 1 month supply, so that compliance was reconciled at follow-up visits, and recorded in accountability logs. Subjects were instructed to take medication with food, (morning and at dinnertime). If subjects missed a dose, they were instructed to resume their normal dose at the next scheduled time, and not to take an extra dose at their next dosing interval if they previously miss a dose.
- Placebo: The placebo is an inert product that looks like a pill and is identical to dimethyl fumarate capsules, but it contains no medicine. Subjects randomized to placebo will be instructed to take placebo twice a day with breakfast and dinner for a period of 4 months.
  Placebo: Placebo capsules were dispensed during routine study appointments. Placebo were dispensed in 1 month supply, so that compliance can be reconciled at monthly follow-up visits, and recorded in accountability logs. Subjects were instructed to take the placebo with food, in the morning and at dinnertime. If subjects missed a dose, they were instructed to resume their normal dose at the next scheduled time, and not to take an extra dose at their next dosing interval if they previously missed a dose.
Arm/Group | Dimethyl Fumarate (Tecfidera®) Capsules | Placebo
Number analyzed (Participants) | 34 | 13
picograms/milliliter (log-transformed)
  Interleukin-6 | 0.038 (0.249) | -0.015 (0.096)
  Tissue necrosis factor-alpha | -0.002 (0.171) | 0.003 (0.257)
  Interleukin-10 | 0.084 (0.253) | -0.036 (0.170)
  Monocyte chemoattractant protein-1 | 0.005 (0.136) | 0.057 (0.157)

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were captured at each visit beginning with Month 1 visit and ending with the Month 5 follow-up visit.
Arm/Group | Dimethyl Fumarate (Tecfidera®) Capsules | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/21
Other Adverse Events (participants affected / at risk) | 27/44 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dimethyl Fumarate (Tecfidera®) Capsules (N=44) | Placebo (N=21)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dimethyl Fumarate (Tecfidera®) Capsules (N=44) | Placebo (N=21)
Flushing (Skin and subcutaneous tissue disorders) | 23 (27) | 0 (0)
Indigestion (Gastrointestinal disorders) | 2 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Cold (Infections and infestations) | 3 (4) | 3 (3)
Sinus Infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes